# **Statistical Analysis Plan (SAP)**

# HISTORI – Home-Based Intervention with Semaglutide Treatment of neuroleptics-related prediabetes

N. Uhrenholt<sup>1,5</sup>, A. Ganeshalingam<sup>2,5</sup>, S. Arnfred<sup>3</sup>, J. Frystyk<sup>2</sup>, P. Gæde<sup>4</sup>, N. Bilenberg<sup>5</sup>

#### **PRIMARY PUBLICATION**

Change in HbA1c, metabolic measures, PANSS and SF-36.

#### **SECONDARY PUBLICATIONS**

- Changes in PANSS Mediators Impact of Weight on Quality of Life-Lite (IWQOL-lite), Medication Adherence Rating Scale (MARS) and weight.
- Changes in cardiovascular risk markers and CAN assessment
- Changes in NAF PET CT scans and body composition.
- Changes in SF-36 Mediators Weight and Simple Physical Activity Questionnaire (SOMPAQ).
- Cost-utility analysis and Cost-effectiveness analysis.
- Insulin resistance a driving factor for prediabetes, dyslipidemia and elevated cardiovascular risk markers?

<sup>&</sup>lt;sup>1</sup>Psychiatry West, Region Zealand, Research Unit West, Slagelse, Denmark.

<sup>&</sup>lt;sup>2</sup>Odense University Hospital, Department of Endocrinology M / Steno Diabetes Centre Odense (SDCO), Odense, Denmark.

<sup>&</sup>lt;sup>3</sup>Psychiatric Research Unit, Copenhagen University Hospital – Psychiatry Region Zealand, Slagelse, Denmark.

<sup>&</sup>lt;sup>4</sup>Næstved, Slagelse og Ringsted Hospital, Department of cardiology and endocrinology, Slagelse, Denmark.

<sup>&</sup>lt;sup>5</sup>Mental Health Services in the Region of Southern Denmark, Child and Adolescent Psychiatry Odense, Odense C, Denmark.

#### **INTRODUCTION**

This document specifies the planned statistical analysis for the RCT-study "HISTORI – Home-Based Intervention with Semaglutide Treatment of neuroleptics-Related prediabetes"

" as carried out following the protocol published in BMJ Open: <a href="https://doi.org/10.1136/bmjopen-2023-077173">https://doi.org/10.1136/bmjopen-2023-077173</a>, and in ClinicalTrials.gov ID NCT05193578

#### TRIAL DESIGN

A two-armed, multi-center, superiority, double-blinded, randomized trial investigating the effect of weekly injections of Semaglutide vs placebo. Each patient will be included in 30 weeks of treatment with weekly injection of Semaglutide 1.34 mg/ml (1 mg) or placebo. The treatment group will start at 0.25 mg Semaglutide per week for 4 weeks, then 0.5 mg per week for 4 weeks. The patients will remain at the highest tolerated dose. There is a 6 week lasting wash-out period for registration of side-effects after each last patient last visit. Setting: Mental health facilities in Region of Southern Denmark and Region of Zealand, Denmark.

#### **RANDOMIZATION**

Randomization 1:1 to Semaglutide or placebo. Block randomization including blocks of either 4 or 6 randomization numbers will be used, and the randomization list will be provided by the manufacturer of Semaglutide and placebo.

#### SAMPLE SIZE

#### PRIMARY OUTCOME (HBA1C CHANGE)

The study requires 154 participants, including an expected 15% dropout. If we conservatively assume that 30 weeks of Semaglutide reduces HbA1c by 0.2%, and that SD equals 0.35%, 65 subjects in each arm are required to obtain a power of 90%, using a 2-sided significance level of 5%.

#### FRAMEWORK

The trial has been designed to investigate whether the new treatment being tested is superior to placebo in terms of efficacy and other relevant outcomes.

#### STATISTICAL INTERIM ANALYSES

Early Identification of Safety Concerns: Monitoring safety outcomes during interim analyses allows for early detection of potential safety issues associated with the treatment. The analysis will be performed blinded through serious adverse events (SAE) and suspected unexpected serious adverse reaction (SUSAR) registrations.

#### TIMING OF FINAL ANALYSIS

All outcomes will be analyzed collectively when all participants have completed the study and when the researchers are still blinded.

#### **SECTION 4: STATISTICAL PRINCIPLES**

#### CONFIDENCE INTERVALS AND P VALUES

Statistical tests will be conducted as two-sided tests with a 5% significance level and a confidence interval of 95%.

#### 1. Holm's Method:

- A step-down procedure that adjusts p-values in a sequential manner.
- It maintains strong control over the family-wise error rate (probability of making one or more Type I errors).

#### ADHERENCE AND PROTOCOL DEVIATIONS

Adherence to the intervention will be measured once weekly. Every pen of semaglutid/placebo has a specific number. Every week, the participants will have to inform the research staff of that number. The number will be inputted in the eCRF. Researchers can then track if the correct numbers are being reported. Furthermore, pens will be collected and checked to see if there are any medicine/placebo left.

Adherence to the intervention will be presented as number of weeks of injections completed. Not completing an injection or a questionnaire or measurement will be defined as a protocol deviation. Major protocol deviations will be summarized. Missing injections or missing data at baseline, week 15 and week 30.

#### ANALYSIS POPULATIONS

Analyses will be performed as intention-to-treat.

PLANNED ANALYSES FOR PRIMARY PUBLICATION: CHANGE IN HBA1C, METABOLIC MEASURES, PANSS AND SF-36

Primary outcome: Main analysis

HbA1c mmol/mol measured at baseline, week 15 and week 30.

#### SECONDARY OUTCOMES TO BE INCLUDED IN THE PRIMARY PUBLICATION

#### Secondary outcomes

- Positive and Negative syndrome scale (PANSS-6), the 36-Item Short Form Health Survey questionnaire (SF-36v2)
- Weight, BMI, Waist Circumference
- Biochemical screening at baseline and after 30 weeks: FBG, FBI, TG, LDL, HDL, C-peptide (proinsulin), liver and renal function test, hemoglobin, amylase and calcium, SHBG, testosterone, FSH, LH, uric acid, hs-CRP and choriogonadotropin (hCG) in all female participants.

#### **SAFETY OUTCOMES**

- Death all causes
- SAE
- GI symptoms
- Worsening of psychiatric symptoms
- Changes in liver function and kidney function

#### PLANNED TABLES AND FIGURES AND CORRESPONDING ANALYSES

Characteristics (as listed in Table 1 below, numerical characteristics marked with [numerical]) of patients at baseline will be reported separately for the two treatment groups.

- Clinical results that align with the normal distribution will be presented as mean with SE, SD or two-sided 95%
   CI.
- Clinical results that do not align with a normal distribution will be presented as median, and 25 and 75 percentile.

Beside the descriptive tables spaghetti and margins plot will be constructed to graphically assess how the parametrization of our model has to be for the primary analysis.

Mixed-effects linear models will be employed to assess the association between the treatment groups and the primary outcome (HbA1c) over time (baseline, week 15 and 30 weeks). These models efficiently handle missing values using the maximum likelihood estimator, assuming the dropout mechanism is missing at random (MAR). The models will include a random intercept per participant. The necessity of a random slope will be evaluated for each model using F-test, and it will be included if it significantly improves the model. In order to test whether the intervention has a statistically significant effect we will employ a likelihood ratio test and use G-estimation where the Q-model will be the mixed effect model to effectively estimate the overall effect size across all timepoints.

In relation to the secondary analysis we will again use the G-estimation framework. For the secondary analysis of PANSS-6 and SF-36 we will use the beta binomial regression as the Q-model and again employ likelihood ratio test to assess whether our intervention has an effect on our secondary outcomes. In relation to weight we will either employ mixed effect model or mixed effect gamma model and again use G-estimation to get interpretable effect sizes.

For the G-estimation approaches we will estimate the confidence intervals by way of bootstrap.

No adjustments for multiple testing will be carried out in Table 1 and no effect sizes for differences between groups will be estimated. Missing observations will be excluded from tests in Table 1, and number for missing observations in each group will be specified.

04-07-2024 Version 1.2

Sample template for the CONSORT diagram showing the flow of participants through each stage of a randomized trial. The text boxes can be modified by clicking on them.



Baseline Table 1 Active Placebo P-value

Age, mean (SD), Years

Female, No. (%)

**Fasting Blood Glucose** 

Smoking no. (%) Alcohol consumptions > 14 units weekly. Diagnosis, No. (%) Schizophrenia Schizotypal disorder Schizoaffective disorder Duration of diagnosis, months, No(%) 6-12 months 12-24 months >24 months Treatment, No. (%) Quetiapine Olanzapine Risperidone **Ziprasidone Paliperidone Aripiprazole** Clozapine Other 1 Drug 2 drugs 3+ drugs **Psychiatric evaluations PANSS-6 Score Positive Score Negative Score SF 36 Physical Component Summary Mental Component Summary** Clinical characteristics, mean (SD) Body weight, kg Waist circumference, cm **BMI** Systolic Blood pressure, mm HG Diastolic Blood pressure, mm HG **Glucose Metabolism** HbA1C, mmol/mol, mean (SD)

| Fasting C-peptide Fasting insulin level Organ function Creatinine Levels ALAT Amylase BASP Bilirubin Cholesterol Level Total LDL HDL Triglycerides Other biochemical variables Testosterone SHBG Urate CRP | |
|---|---|
| Organ function Creatinine Levels ALAT Amylase BASP Bilirubin Cholesterol Level Total LDL HDL Triglycerides Other biochemical variables Testosterone SHBG Urate | Fasting C-peptide |
| Creatinine Levels ALAT Amylase BASP Bilirubin Cholesterol Level Total LDL HDL Triglycerides Other biochemical variables Testosterone SHBG Urate | Fasting insulin level |
| ALAT Amylase BASP Bilirubin Cholesterol Level Total LDL HDL Triglycerides Other biochemical variables Testosterone SHBG Urate | Organ function |
| Amylase BASP Bilirubin Cholesterol Level Total LDL HDL Triglycerides Other biochemical variables Testosterone SHBG Urate | Creatinine Levels |
| BASP Bilirubin Cholesterol Level Total LDL HDL Triglycerides Other biochemical variables Testosterone SHBG Urate | ALAT |
| Bilirubin Cholesterol Level Total LDL HDL Triglycerides Other biochemical variables Testosterone SHBG Urate | Amylase |
| Cholesterol Level Total LDL HDL Triglycerides Other biochemical variables Testosterone SHBG Urate | BASP |
| Total LDL HDL Triglycerides Other biochemical variables Testosterone SHBG Urate | Bilirubin |
| LDL HDL Triglycerides Other biochemical variables Testosterone SHBG Urate | Cholesterol Level |
| HDL Triglycerides Other biochemical variables Testosterone SHBG Urate | Total |
| Triglycerides Other biochemical variables Testosterone SHBG Urate | LDL |
| Other biochemical variables Testosterone SHBG Urate | HDL |
| Testosterone SHBG Urate | Triglycerides |
| SHBG Urate | Other biochemical variables |
| Urate | Testosterone |
| | SHBG |
| CRP | Urate |
| | CRP |

# PRIMARY OUTCOME AND SECONDARY OUTCOMES

Table 2: Changes in endpoints from baseline to week 30.

Variables Active Placebo Estimated P-value difference

## **Glucose Metabolism**

Hemoglobin

HbA1C, mmol/mol, mean (SD)

**Fasting Blood Glucose** 

**Fasting C-peptide** 

Fasting insulin level

**PANSS Score** 

**Positive** 

| Ne | gat | iv€ | • |
|----|-----|-----|---|

Physical Component Summary

SF - 36

**Mental Component Summary** 

Clinical characteristics, mean (SD)

Body weight, kg

Waist circumference, cm

вмі

Systolic Blood pressure, mmHg

Diastolic Blood pressure,

mmHg

**Organ function** 

**Creatinine Levels** 

ALAT

**Amylase** 

**BASP** 

**Bilirubin** 

**Cholesterol Level** 

Total

LDL

HDL

**Triglycerides** 

Other biochemical variables

**Testosterone** 

**SHBG** 

Urate

**CRP** 

Hemoglobin

| Table 3. Char | Changes after 15 and 30 weeks treatment with Semaglutide or placebo | | | |
|---|---|---|---|---|
| | | 21 1 1 1 1 2 | | 2./.1 |
| | Active - Week 15 | Placebo- Week 15 | Mean difference | P-Value |
| HbA1c | | | | |
| PANSS | | | | |
| SF-36 | | | | |
| Weight | | | | |
| | Active - end of study | Placebo - end of study | Mean difference | P-Value |
| HbA1c | | | | |
| PANSS | | | | |
| SF-36 | | | | |
| Weight | | | | |

HbA1c mol/mmol, PANSS and SF-36 are numerical values and weight Kg. Values are represented as number (%). p Values were obtained from chi square test.





 ${\bf Blue: Placebo.\ Orange: Semaglutide.}$ 



#### **SAFETY OUTCOMES**

Severe safety outcomes will be reported in table 3.

Variables Active Placebo Estimated P-value difference

#### **SERIOUS ADVERSE EVENTS**

Death

Hopitalisation

Somatic illness

Hypoglycemia

**Psychiatric illness** 

Admission – worsening of schizophrenia

Voluntarily institutional care

| Comp | ulsory | / institutional | care |
|------|--------|-----------------|------|

Expected adverse events and side effects will be reported table 4

Variables Active Placebo **Estimated** P-value difference **Side effects** Nausea Diarrhea **Abdominal pain** Dyspepsia **Flatulence** Constipation Vomiting **Other Adverse events Fatigue** Headache Dizziness Infections Flue like symptoms **Pneumonia Abdominal infection Urinal Tract infections Biochemical safety** Change in liver function **Change in Kidney** 

**Elevated Amylase levels** 

function

Smoking no. (%)

PLANNED ANALYSES FOR SECONDARY PUBLICATION: CHANGES IN PANSS – MEDIATORS - IMPACT OF WEIGHT ON QUALITY OF LIFE-LITE (IWQOL-LITE), MEDICATION ADHERENCE RATING SCALE (MARS) AND WEIGHT.

Characteristics (as listed in Table 1 below, numerical characteristics marked with [numerical]) of patients at baseline will be reported separately for the two treatment groups.

- Clinical results that align with the normal distribution will be presented as mean with SE, SD or two-sided 95%
   CI.
- Clinical results that do not align with a normal distribution will be presented as median, and 25 and 75 percentile.

Beside the descriptive tables spaghetti and margins plot will be constructed to graphically assess how the parametrization of our model must be for the primary analysis.

The primary analysis will utilize the G-estimation framework. The Q-model in this regard will be a structural equation model where the longitudinal aspect and effect modification will be incorporated into the framework. A directed acyclic graphs will be constructed to visualize which assumption we have made concerning the underlying causal structure. For the G-estimation approaches we will estimate the confidence intervals by way of bootstrap.

No adjustments for multiple testing will be carried out in Table 1 and no effect sizes for differences between groups will be estimated. Missing observations will be excluded from tests in Table 1, and number for missing observations in each group will be specified.

## PLANNED ANALYSES SECONDARY PUBLICATION:. CHANGES IN CAN ASSESSMENT

| Baseline Tabel 1 | Active | Placebo | P-value |
|-----------------------|--------|---------|---------|
| Age, mean (SD), Years | | | |
| Female, No. (%) | | | |

| Alcohol consumptions > 14 units weekly. |
|-----------------------------------------|
| Diagnosis, No. (%) |
| Schizophrenia |
| Schizotypal disorder |
| Schizoaffective disorder |
| Duration of diagnosis, months, No (%) |
| 6-12 months |
| 12-24 months |
| >24 months |
| Treatment, No. (%) |
| Quetiapine |
| Olanzapine |
| Risperidone |
| Ziprasidone |
| Paliperidone |
| Aripiprazole |
| Clozapine |
| Other |
| Psychiatric evaluations |
| PANSS-6 Score |
| P1 |
| P2 |
| P3 |
| N1 |
| N4 |
| N6 |
| Clinical characteristics, mean (SD) |
| Body weight, kg |
| Waist circumference, cm |
| вмі |
| Systolic Blood pressure, mmHg |
| Diastolic Blood pressure, mmHg |
| Glucose Metabolism |
| HbA1C, mmol/mol, mean (SD) |
| Fasting Blood Glucose |
| Fasting C-peptide |
| Fasting insulin level |

| Organ function |
|-----------------------------|
| Creatinine Levels |
| ALAT |
| Amylase |
| BASP |
| Bilirubin |
| Cholesterol Level |
| Total |
| LDL |
| HDL |
| Triglycerides |
| Other biochemical variables |
| Testosterone |
| SHBG |
| Urate |
| CRP |
| Hemoglobin |

| | Schizophrenia | Healthy control | P-value |
|---|---|---|---|
| Degree of CAN | | | |
| No diagnosis of CAN, n/N (%) | | | |
| Early CAN, n/N (%) | | | |
| Manifest CAN, n/N (%) | | | |
| | Schizophrenia | Diabetes mellitus type 2 | |
| Degree of CAN | | | |
| No diagnosis of CAN, n/N (%) | | | |
| Early CAN, n/N (%) | | | |
| Manifest CAN, n/N (%) | | | |



| Table 3. Prevalence of CAN among patients with schizophrenia in various Antipsychotic treatment | | | |
|---|---|---|---|
| | No diagnosis of CAN, n/N (%) | Early CAN, n/N (%) | Manifest CAN, n/N (%) |
| Olanzapine | | | |
| Quetiapine | | | |
| Risperidone | | | |
| Ziprasiode | | | |
| Palliperidone | | | |
| Aripiprazole | | | |
| Clozapine | | | |
| Other | | | |
| CAN: cardiovascular autonoi | mic neuropathy. Values are represented as n | umber (%). | |
| p Values were obtained from | n chi square test. | | |

| Table 4. Changes in CAN after week | s treatment with Semaglutide o | or placebo | |
|---|---|---|---|
| | Active - baseline | Placebo- baseline | P-value |
| Degree of CAN | | | |
| No diagnosis of CAN, n/N (%) | | | |
| Early CAN, n/N (%) | | | |
| Manifest CAN, n/N (%) | | | |
| | Active - end of study | Placebo - end of study | |
| Degree of CAN | | | |
| No diagnosis of CAN, n/N (%) | | | |
| Early CAN, n/N (%) | | | |
| Manifest CAN, n/N (%) | | | |
| CAN: cardiovascular autonomic neu | ropathy. Values are represente | ed as number (%). | |
| p Values were obtained from chi so | juare test. | | |

PLANNED ANALYSES SECONDARY PUBLICATION: CHANGES IN NAF PET CT SCANS AND BODY COMPOSITION – A PILOT STUDY IN PROJECT HISTORI

| Baseline Tabel 1 | Active | Placebo | P-value |
|-----------------------------------------|--------|---------|---------|
| Age, mean (SD), Years | | | |
| Female, No. (%) | | | |
| Smoking no. (%) | | | |
| Alcohol consumptions > 14 units weekly. | | | |
| Diagnosis, No. (%) | | | |
| Schizophrenia | | | |
| Schizotypal disorder | | | |
| Schizoaffective disorder | | | |
| Duration of diagnosis, months, No(%) | | | |
| 6-12 months | | | |
| 12-24 months | | | |
| >24 months | | | |
| Treatment, No. (%) | | | |
| Quetiapine | | | |
| Olanzapine | | | |
| Risperidone | | | |
| Ziprasidone | | | |
| Paliperidone | | | |
| Aripiprazole | | | |
| Clozapine | | | |
| Other | | | |

| Psychiatric evaluations |
|-------------------------------------|
| PANSS-6 Score |
| P1 |
| P2 |
| P3 |
| N1 |
| N4 |
| N6 |
| Clinical characteristics, mean (SD) |
| Body weight, kg |
| Waist circumference, cm |
| вмі |
| Systolic Blood pressure, mmHg |
| Diastolic Blood pressure, mmHg |
| Glucose Metabolism |
| HbA1C, mmol/mol, mean (SD) |
| Fasting Blood Glucose |
| Fasting C-peptide |
| Fasting insulin level |
| Organ function |
| Creatinine Levels |
| ALAT |
| Amylase |
| BASP |
| Bilirubin |
| Cholesterol Level |
| Total |
| LDL |
| HDL |
| Triglycerides |
| Other biochemical variables |
| Testosterone |
| SHBG |
| Urate |
| CRP |
| Hemoglobin |

| Table 2. NAF uptake in healthy population and study population | | | |
|---|---|---|---|
| | Non schizophrenic population | Study population | P-value |
| NAF uptake Total | | | |
| NAF uptake BMI 27 - 30 | | | |
| NAF uptake BMI 30 - 40 | | | |
| NAF uptake BMI 40+ | | | |
| NAF: Sodiumflouride uptake. | Values are represented as number (%). | | |
| p Values were obtained from chi square test. | | | |

| | Active - baseline | Placebo- baseline | P-value |
|---|---|---|---|
| NAF uptake Total | | | |
| NAF uptake BMI 27 - 30 | | | |
| NAF uptake BMI 30 - 40 | | | |
| NAF uptake BMI 40+ | | | |
| | Active - end of study | Placebo - end of study | |
| NAF uptake Total | | | |
| NAF uptake BMI 27 - 30 | | | |
| NAF uptake BMI 30 - 40 | | | |
| NAF uptake BMI 40+ | | | |









| Baseline Tabel 5 | Active | Placebo | P-value |
|---------------------|--------|---------|---------|
| Adiponectin | | | |
| TNF-alfa | | | |
| IL-6 | | | |
| <b>Leptin</b> | | | |
| IGF-1 | | | |
| GDF-15 | | | |
| NT ProBNP | | | |
| <b>Homocysteine</b> | | | |
| <b>Fibrinogen</b> | | | |
| Lp(a) | | | |
| ApoB | | | |

PLANNED ANALYSES SECONDARY PUBLICATION: CHANGES IN SF-36 - MEDIATORS - WEIGHT AND SIMPLE PHYSICAL ACTIVITY QUESTIONNAIRE (SOMPAQ).

See analysis plan for PANSS mediators. The same statistical approach will be applied.

# IS INSULIN RESISTANCE A KEY DRIVING FACTOR FOR PREDIABETES, DYSLIPIDEMIA AND ELEVATED CARDIOVASCULAR RISK MARKERS?

| Baseline Tabel 1 | Active | Placebo | P-value |
|-----------------------------------------|--------|---------|---------|
| Age, mean (SD), Years | | | |
| Female, No. (%) | | | |
| Smoking no. (%) | | | |
| Alcohol consumptions > 14 units weekly. | | | |
| Diagnosis, No. (%) | | | |
| Schizophrenia | | | |
| Schizotypal disorder | | | |
| Schizoaffective disorder | | | |
| Duration of diagnosis, months, No(%) | | | |
| 6-12 months | | | |
| 12-24 months | | | |
| >24 months | | | |
| Treatment, No. (%) | | | |
| Quetiapine | | | |
| Olanzapine | | | |
| Risperidone | | | |
| Ziprasidone | | | |
| Paliperidone | | | |
| Aripiprazole | | | |
| Clozapine | | | |
| Other | | | |
| Psychiatric evaluations | | | |
| PANSS-6 Score | | | |
| P1 | | | |
| P2 | | | |
| Р3 | | | |
| N1 | | | |
| N4 | | | |
| N6 | | | |
| Clinical characteristics, mean (SD) | | | |
| Body weight, kg | | | |

Waist circumference, cm BMI Systolic Blood pressure, mmHg Diastolic Blood pressure, mmHg **Glucose Metabolism** HbA1C, mmol/mol, mean (SD) **Fasting Blood Glucose Fasting C-peptide** Fasting insulin level **Organ function Creatinine Levels** ALAT **Amylase BASP Bilirubin Cholesterol Level Total** LDL HDL **Triglycerides** Other biochemical variables **Testosterone SHBG** 

Baseline Tabel 2 Active Placebo P-value

HOMA-2B

Urate CRP Hemoglobin

**HOMA2S** 





Mediator analysis





Alternative for table 3 for PRIMARY OUTCOME (HBA1C CHANGE)

| | Active - Week 15 | Placebo - Week 15 | Mean<br>difference | P-value |
|---|---|---|---|---|
| HbA1c | | | | |
| PANSS-6 | | | | |
| SF-36 | | | | |
| Weight | | | | |
| | Active - end of study | Placebo - end of study | Mean<br>difference | P-value |
| HbA1c | | | | |
| PANSS-6 | | | | |
| SF-36 | | | | |
| Weight | | | | |
| | Active - marginal | Placebo - marginal | Mean<br>difference | P-value |
| HbA1c | | | | |
| PANSS-6 | | | | |
| SF-36 | | | | |
| Weight | | | | |
| | HbA1c mol/mmol, PANSS-6 and SF-36 are numerical values and weight is | | | |
| measured | l in Kg. The p-values | are either based on the | e z or likelihood r | atio test. |

NCT05193578 Unique Protocol ID: Eudra CT 2020-004374-22

4<sup>th</sup> of July 2024 Version 1.0

Two different conclusions before unblinding. Treatment A vs. B.

Home-based Intervention With Semaglutide Treatment Of Neuroleptica-Related Prediabetes

# Treatment A is the investigated drug.

Patients receiving investigated drug Semaglutide (group A) demonstrate significant reductions in HbA1c at week 15 and week 30, when compared to patients receiving placebo (group B). Cases of pre-diabetes were reduced in group A compared to group B. Both findings are clinically meaningful and provide evidence that Semaglutide can normalize glucose levels in patients with schizophrenia and prediabetes. Furthermore, patients receiving Semaglutide reported superior physical health status compared to patients receiving placebo at both week 15 and week 30. Thus, Semaglutide also improves patients' experience of their physical health. In contrast, there were no differences between the two interventions in self-reported mental health status or positive and negative symptoms of schizophrenia. In conclusion, we recommend treatment with Semaglutide for patients with schizophrenia and prediabetes.

# Treatment B is the investigated drug.

Patients receiving investigated drug Semaglutide (group B) demonstrate significantly higher levels of HbA1c at week 15 or week 30, when compared to patients receiving treatment with placebo (group A). Reduction in cases with prediabetes were also less in patients receiving Semaglutide (group B). Differences are clinically meaningful and this provides evidence that Semaglutide is inferior to placebo in normalizing glucose levels in patents with schizophrenia and prediabetes. Furthermore, patients receiving Semaglutide reported inferior physical health status compared to the placebo group. In contrast, there were no differences between the two interventions in self-reported mental health status or positive and negative symptoms of schizophrenia. In conclusion, we cannot recommend treatment with Semaglutide for patients with schizophrenia and prediabetes.